CLINICAL TRIAL: NCT04482660
Title: Characterization of Cerebral Tau Aggregates With 18F-RO6958948 PET in the ALFA Population
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Collaborators: Hoffmann-La Roche (Industry); Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: tau-PET/BBRC2019
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET (Experimental)
  Interventions: Procedure: Positron emission tomography with 18F-RO6958948

INTERVENTIONS:
Procedure: Positron emission tomography with 18F-RO6958948 — tau PET ()

SUMMARY:
This study will characterize tau tracer retention by Positron Emission Tomography (PET) as a function of amyloid levels transversally and longitudinally.

DETAILED DESCRIPTION:
CROSS-SECTIONAL OBJECTIVES

* To measure 18F-RO6958948 retention in selected participants of ALFA-related studies as a function of amyloid levels.
* To study the relation between 18F-RO6958948 retention and amyloid levels.
* To characterize imaging correlates as a function of tau and amyloid levels.
* To study the role of tau retention on cognitive performance.
* To define predictors of tau retention.

LONGITUDINAL OBJECTIVES

* To measure tau accumulation and spreading in participants of the ALFA-related studies of BBRC as a function of baseline amyloid levels.
* To study the dynamic relation between tau spreading and amyloid levels longitudinally.
* To define predictors of tau spreading.

ELIGIBILITY:
Inclusion Criteria:

1. To sign the study informed consent form approved by the corresponding authorities.
2. Men and women that have participated in a BBRC-sponsored study, including the ALFA project (STUDY 45-65 FPM/2012), the ALFA+ cohort study (ALFA - FPM - 0311), the ALFA cognition study (ALFAcognition/BBRC2017) or the BarcelonaBeta Dementia Prevention Research Clinic study (BBRC-DemPrev-2018).
3. Participants with an available cerebral MRI within the last 12 months not suggestive of radiological incidental findings constituting an exclusion criterion.
4. Known cognitive status based on the cognitive workup of the BBRC-sponsored studies specified above. Cognitive status should have been determined within the last 12 months.
5. Known AB and tau status.
6. Good knowledge of the language and being literate.
7. Female participants should be post-menopausal or present a negative pregnancy test at the moment of PET acquisition.

Exclusion Criteria:

1. Presence of clinically relevant psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria: major depressive disorder, generalized anxiety disorder, schizophrenia and bipolar disorder, as assessed in the BBRC-sponsored studies specified above.
2. Participants with visual and/or hearing impairment.
3. History of encephalitis, ictus or seizures excluding feverish convulsions during childhood, as assessed in the BBRC-sponsored studies specified above.
4. Severe cerebral macrovascular (i.e., multi-stroke) disease or brain tumour (metastasis/brain cancer) as verified by MRI.
5. Previous participation in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening and/or administration of a radiopharmaceutical within 10 radioactive half-lives prior to study drug administration in this study.
6. Clinically relevant renal or hepatic insufficiency.
7. Any other clinically important condition that may jeopardize the study or be dangerous for the participant.
8. Active drug or alcohol abuse, as assessed in the BBRC-sponsored studies specified above.
9. Previous intolerance to PET studies or known hypersensitivity to 18F-RO6958948.
10. Being pregnant or breast-feeding.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cerebral tau positivity | at inclusion
  Prevalence of cerebral tau positivity assessed by 18F-RO6958948 PET
tau accumulation and spreading | 2 years
  To predictors of tau spreading

CONTACTS AND LOCATIONS:
Locations (1):
- BarcelonaBeta Brain Research Center, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No